CLINICAL TRIAL: NCT07392801
Title: Study of Advanced Glycation End-products Accumulation in Patients Under Long-Term Parenteral Nutrition (NUPARAGE2)
Brief Title: AGE Accumulation in Patients on Long-term Parenteral Nutrition (NUPARAGE2)
Acronym: NUPARAGE2
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2025/048
Record Dates: First submitted 2026-01-29; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Chronic Intestinal Insufficiency; Advanced Glycation and Products; Parenteral Nutrition
Keywords: parenteral nutrition; Advanced Glycation End Products; Oxidative Stress; Metabolic Diseases; Cardiovascular Diseases; Short Bowel Syndrome; chronic intestinal insufficiency
MeSH Terms: conditions — Hyperphagia; Metabolic Diseases; Cardiovascular Diseases; Short Bowel Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients starting long-term parenteral nutrition (Other): Observational follow-up of patients starting long-term parenteral nutrition
  Interventions: Other: Non-invasive skin AGE measurements

INTERVENTIONS:
Other: Non-invasive skin AGE measurements — Non-invasive skin AGE measurements at baseline, 6 and 12 months; collection and analysis of parenteral nutrition bag samples; routine metabolic assessments; dietary records, glucose holter, plasma glycated hemoglobin and fructosamine assays.

SUMMARY:
This prospective and observational study aims to evaluate the accumulation of advanced glycation end-products (AGEs) in adult and pediatric patients starting long-term parenteral nutrition, by non-invasive skin AGE measurements over a 12-month follow-up.

DETAILED DESCRIPTION:
Advanced Glycation End-products (AGEs) result from non-enzymatic glycation of proteins, lipids, or amino acids, and accumulate progressively with age, hyperglycemia, and oxidative stress. Their accumulation is associated with metabolic and cardiovascular complications in chronic diseases. Preliminary data suggest that patients on long-term parenteral nutrition may experience increased AGE accumulation due to high intravenous glucose exposure. However, prospective data evaluating AGE kinetics from the initiation of parenteral nutrition are lacking.

Skin AGE levels will be measured non-invasively at baseline, 6 months, and 12 months using the AGE Reader© device. Nutrition bag samples will be analyzed for AGE content via HPLC-MS.

Patients will be monitored during routine consultations every 6 months. Biological metabolic parameters (HbA1c, fructosamine, lipid profile), nutritional data, and 3-day dietary records will be collected at each time point. Samples from parenteral nutrition bags will be frozen at -20°C or colder and analyzed centrally after the last patient visit.

ELIGIBILITY:
Inclusion Criteria:

* Patients (adults and children, all ages) initiating long-term parenteral nutrition
* Followed at CHU de Bordeaux or Robert Debré Hospital (APHP)
* Covered by French Social Security system
* Written informed consent obtained from patient (if adult) or legal guardian (if minor)

Exclusion Criteria:

* Fitzpatrick skin type ≥ V (darker skin tones)
* Forearm tattoos at the site of measurement
* For patients included under 1 year of age: patients born prematurely (before 37 weeks of amenorrhea)
* Pregnant or breastfeeding women.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Skin AGE levels | Baseline, 12 months
  Change in skin AGE levels between baseline and 12 months after initiation of parenteral nutrition (Visit M12).

SECONDARY OUTCOMES:
Advanced Glycation End-products | 6 months
  Compare skin AGE (Advanced Glycation End-products) levels with Age levels in parenteral nutrition bags (M6)
Risk factors | Baseline, 6 months and 12 months
  Search for risk factors for AGE accumulation linked to dietary habits
Skin AGE and metabolic/cardiovascular status | Baseline, 6 months and 12 months
  To investigate whether there is an association between skin AGE levels and the metabolic and cardiovascular status of patients.
AGE and hyperglycaemic episodes | Baseline, 6 months and 12 months
  To investigate whether there is an association between skin AGE levels and the number, duration and intensity of hyperglycaemic episodes during parenteral nutrition infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Florian POULLENOT, MD, Principal Investigator — University Hospital, Bordeaux
Locations (3):
- France (3):
  - CHU de Bordeaux-Hôpital des enfants GH Pellegrin, Bordeaux
  - AP-HP - Hopital Robert Debré, Paris
  - CHU de Bordeaux - Hôpital Haut Lévêque, Pessac